CLINICAL TRIAL: NCT07080645
Title: Biosilicate as a Desensitizing Agent in Teeth With Molar Incisor Hypomineralization in Children: A Randomized Clinical Trial
Brief Title: BIOSILITACE AS A DESENSITIZING AGENTIN HMI
Acronym: BDAHMI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Paulla Iaddia Zarpellon Barbosa, PESQUISADOR, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIOSILIC2025; BIOSILC HMI (Other: CNPQ)
Record Dates: First submitted 2025-04-02; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Sensitive Dentin; Hypomineralization Molar Incisor; Pain
Keywords: pain; Molar-Incisor Hypomineralization; biosilicate; dentin hypersensitivity; tooth enamel; child
MeSH Terms: conditions — Dentin Sensitivity; Molar Hypomineralization; Pain | interventions — Analgesia; sodium oxide-calcium oxide-silicon dioxide-diphosphorus pentoxide; Fluoride Treatment

STUDY DESIGN:
Intervention Model Description: According to the sample calculation of this study, 42 children (21 per group) will be selected, who have teeth with Molar-Incisor Hypomineralization and painful sensitivity in those teeth, recruited from Municipal Schools in Ribeirão Preto, São Paulo, Brazil, and children treated at the Pediatric Dentistry Clinic and the Dental Enamel Clinic of FORP USP. The children included in the study will be subdivided into three randomized treatment options, which are: Group 1: Fluoridated varnish (Duraphat® Colgate, Brazil); Group 2: Biosilicate® 10%. The randomization sequence will be generated using the envelope method. A numerical sequence (1 and 2) will be printed, which will correspond sequentially to the three groups (GI and GII).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To ensure the first stage of blinding in the study, the patient will not know which group and type of treatment the tooth will receive. Therefore, we will attempt to standardize some methods to ensure this reliability. The products to be tested will be removed from their original containers and placed in identical 10ml white bottles. The second stage concerns the evaluator. All treatments will be performed by a single operator, and the tests will be applied by another evaluator. In this way, the evaluator will not know the group allocation or the type of intervention that was performed.To increase the reliability of the results, the statistician will also not know the allocation or which groups correspond to each treatment. They will only receive a table with letters representing the groups as A and B and the test values, without knowing which group or interventions were carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biosilicate® 10% (Experimental): Supervised tooth brushing will be performed with fluoride-free toothpaste. Then, the tooth affected by MIH will be cleaned with sterile gauze, isolated with a cotton roll, and subsequently, the operator will apply a solution using a microapplicator to all the free surfaces of the selected teeth. This solution will either be a 10% Biosilicate® solution or fluoride varnish (Duraphat®). All products will be removed from their original containers and placed in identical 10ml plastic bottles, white and standardized. The different products will be applied equally for 15 seconds according to the application protocol. Immediately after application, sensitivity tests will be performed using the SCASS and VAS protocols, and will be repeated 1, 2, 4, and 8 weeks after the completion of the treatment. The form for recording the results for each patient is provided in.
  Biosilicate (Na₂O-CaO-SiO₂-P₂O₅), a finely particulate glass-ceramic with a high degree of crystallinity (~99.5%), exhibiting an
  Interventions: Other: Pain Relieving; Other: topical application
- Duraphat® (Active Comparator): Initially, the child will be instructed not to consume any food or drink for up to 40 minutes after the treatment. Oral hygiene instructions will be given, and a kit with a toothbrush and fluoride toothpaste will be provided. In all groups, the treatment protocols will be applied once a week for 4 consecutive weeks. Supervised tooth brushing will be performed with fluoride-free toothpaste, followed by cleaning the tooth affected by MIH with sterile gauze, isolating it with a cotton roll, and then, the operator will apply a solution to all the free surfaces of the selected teeth using a microapplicator. The solution will either be 10% Biosilicate® solution, fluoride varnish (Duraphat®). All products will be removed from their original containers and placed in identical 10ml plastic bottles, white and standardized. The different products will be applied equally for 15 seconds according to the application protocol.
  Interventions: Other: Pain Relieving; Other: topical application

INTERVENTIONS:
Other: Pain Relieving — aim to relieve tooth pain with HMI Biosilicate
  Other Names: Pain relieving dentin; Dentin Hypersensitivity; Molar-Incisor Hypomineralization and Biosilicate
Other: topical application — the operator will apply a solution to all the free surfaces of the selected teeth using a microapplicator. The solution will either be 10% Biosilicate® solution, fluoride varnish (Duraphat®), or distilled water . All products will be removed from their original containers and placed in identical 10ml plastic bottles, white and standardized. The different products will be applied equally for 15 seconds according to the application protocol.

SUMMARY:
Molar-Incisor Hypomineralization (MIH) is a qualitative enamel defect caused by systemic hypomineralization that affects one to four first permanent molars, and may or may not involve incisors. The clinical repercussions associated with MIH can be characterized by: painful hypersensitivity, post-eruptive fractures, rapid progression of caries lesions in newly erupted first permanent molars, difficulty in achieving effective anesthesia, aesthetic impairments, and patient fear and anxiety. To date, there is no consensus on the best treatment for sensitivity in teeth with MIH, thus managing sensitivity in these teeth remains a significant challenge. The aim of this study is to evaluate the effectiveness of a 10% Biosilicate® solution as a desensitizing agent in MIH teeth in children, compared to Fluoride varnish (Duraphat® Colgate, Brazil). Children aged 6 to 12 years will be selected for this study, with a total of 63 participants diagnosed with MIH, and a sensitivity score ≥2 on the SCASS scale. The children will be randomly divided into two groups (n=21): GI: Duraphat®, GII: Biosilicate®. Interventions will be performed once a week for 4 consecutive weeks, followed by 8 weeks of follow-up. The results will be subjected to statistical tests with a 95% confidence level (α = 0.05).

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of a 10% Biosilicate® solution as a desensitizing agent in MIH teeth in children, compared to Fluoride varnish (Duraphat® Colgate, Brazil). The children included in the study will be subdivided into three randomized treatment options, which are: Group 1: Fluoridated varnish (Duraphat® Colgate, Brazil); Group 2: Biosilicate® 10%. The randomization sequence will be generated using the envelope method. A numerical sequence (1 and 2) will be printed, which will correspond sequentially to the three groups (GI and GII). The numbers will be placed in envelopes with the same characteristics and then sealed. The implementation of the random allocation sequence will be carried out by a single researcher, who will use the previously sealed envelopes along with the numbers corresponding to the treatments to be administered. As each child is included in the study, an envelope will be labeled with the child's name and will only be opened by the operator before the start of the treatment. Children with the potential for inclusion in the research will be referred for clinical examination in the mobile dental unit (Dental Case), and those with at least one first permanent molar affected by MIH and reporting hypersensitivity, with or without structure loss, will be invited to participate. The complaint of sensitivity will be confirmed by applying a 1-second air blast at a distance of 1 centimeter from the occlusal surface of the tooth; a score of 2 or 3 on the Schiff Cold Air Sensitivity Scale (SCASS) will be considered a positive result.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes, aged between 6 and 12 years.
* Children who have at least one first permanent molar with Molar-Incisor Hypomineralization, showing distinct white or cream opacity (score 21), yellowish or brown opacity (score 22), and/or post-eruptive enamel fracture (score 3), and presence of painful sensitivity when stimulated, with a score of 2 or 3 as evaluated using the SCASS scale.
* Children without systemic and/or cognitive impairments.

Exclusion Criteria:

* Previous use of desensitizing therapy in the last 6 months;
* Use of analgesic and anti-inflammatory medications during the previous 3 days;
* Use of orthodontic appliances;
* Teeth with extensive restorative procedures, such as stainless steel crowns, which prevent the assessment of painful sensitivity;
* Teeth with amelogenesis imperfecta or dentinogenesis imperfecta;
* Children with systemic and/or cognitive impairments.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
The Visual Analogue Scale (VAS) | 3 months
  VAS (Visual Analog Scale), a psychometric assessment scale to measure the amount of pain the patient feels, which is reported by the patient himself and can vary from no pain (0) to extreme pain (10).The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best). In some studies, horizontal scales are orientated from right to left, and many investigators use vertical VAS.

SECONDARY OUTCOMES:
Schiff Cold Air Sensitivity Scale (SCASS) | 3 months
  The SCASS is scored as follows: 0 = subject does not respond to the stimulus; 1 = subject does not respond to the stimulus, but considers the stimulus painful; 2 = subject responds to the air stimulus and moves away from the stimulus; and 3 = subject responds to the air stimulus, moves away from the stimulus and requests immediate interruption of the stimulus (Schiff et al., 2009).

CONTACTS AND LOCATIONS:
Overall Officials: doutoranda, Principal Investigator — NÃO FILIADO
Locations (1):
- Faculdade de Odontologia de Ribeirão Preto FORP USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Shrestha R, Upadhaya S, Bajracharya M. Prevalence of molar incisor hypomineralisation among school children in Kavre. Kathmandu Univ Med J (KUMJ). 2014 Jan-Mar;12(45):38-42. doi: 10.3126/kumj.v12i1.13631. PMID 25219992
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38920887/